CLINICAL TRIAL: NCT01101347
Title: A Feasibility Study of the Surpass Aneurysm-Embolization System in Intracranial Arteries
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Product received Approval for Commercial Distribution
Sponsor: Surpass Medical Ltd. (Industry)
Responsible Party: Marc Litzenberg, Surpass Medical, Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-03
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aneurysm-Embolization System (Experimental)
  Interventions: Device: Aneurysm-Embolization System

INTERVENTIONS:
Device: Aneurysm-Embolization System

SUMMARY:
The purpose of this study is to evaluate safety and performance of the Surpass Aneurysm-Embolization System.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the nature of the procedure and provides written informed consent.
* Subject is willing to return to the investigational site for the thirty day and six month follow-up evaluations.
* Age 18 years to 80 years.
* Subject with a non-ruptured saccular, or fusiform intracranial aneurysm arising from a parent vessel with a diameter of > 2mm and < 6mm.

Exclusion Criteria:

* Pregnancy
* Enrollment in another trial
* Allergy or contraindication to aspirin, clopidogrel, heparin, local or general anesthesia
* History of life threatening allergy to contrast dye.
* Major surgery within previous 30 days or planned in the next 90 days after enrollment date.
* Severe neurological deficit that renders the patient incapable of living independently
* Dementia or psychiatric problem that prevents the patient from completing required follow up
* Co-morbid conditions that may limit survival to less than one year
* Subject with anatomy not appropriate for endovascular treatment due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy.
* Subject with an intracranial mass (tumor (except meningioma), abscess, or other infection), or is undergoing radiation therapy for carcinoma or sarcoma of the head or neck region.
* Subject has a history of bleeding diathesis or coagulopathy, international normalized ratio (INR) greater than 1.5, or will refuse blood transfusions.
* Subject has a serum creatinine level greater than 2.0 mg/dL (within 7 days of procedure) which the investigator determines restricts the use of contrast agents.
* Subject has a previously implanted intracranial stent associated with the symptomatic distribution within the past 12 weeks prior to enrollment date
* Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to enrollment date
* Subject has a previously implanted carotid stent associated with the symptomatic distribution within the past 12 weeks prior to enrollment date
* Subject has uncontrolled atrial fibrillation or known cardiac disorders likely to be associated with cardioembolic symptoms.
* Subject had a subarachnoid hemorrhage within 12 weeks prior to the enrollment date.
* Subject with resistance to ASA and/or Clopidogrel.
* Subject with two or more aneurysms in associated distribution - unless the device is used to treat both aneurysms.
* Subject has a non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm.
* Target aneurysm is expected to require more than one device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Gupta, MD, Principal Investigator — Medanta, Medcity